CLINICAL TRIAL: NCT07354997
Title: Research on the Construction and Driving Mechanisms of an Interactive Management Model for Pre-diabetic Patient Groups Based on Virtual Health Communities
Brief Title: Establishing a Virtual Health Community Management Model for Pre-Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiling Hu, Chief Nurse, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG2023-262-03
Record Dates: First submitted 2025-12-15; First posted 2026-01-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-diabetes Virtual Community Experience Group (Experimental)
  Interventions: Other: Pre-diabetes Virtual Community

INTERVENTIONS:
Other: Pre-diabetes Virtual Community — By collecting general information, physical measurements, glucose and lipid metabolism indicators, dietary habits, and exercise routines from prediabetic patients, these details are input into the virtual community programme for prediabetes. The virtual community evaluates the input data, alerts healthcare professionals to patients requiring immediate intervention, and provides guidance for the forthcoming week regarding diet, exercise, and other health aspects (including dietary and exercise advice for prediabetic patients), alongside risk alerts.

SUMMARY:
This study builds upon the previously developed virtual health community platform, aiming to address the group characteristics and psychological traits of prediabetic patients. By employing intervention mapping to construct a group interaction management model, it seeks to develop a mobile platform integrating "gamified knowledge acquisition and motivation", "immersive lifestyle practice experiences", and "sustained community interaction management". The primary focus is on fostering patients' continuous and proactive engagement. Subsequently, a single-arm controlled trial will validate the model's efficacy, aiming to address the health management challenges faced by China's substantial prediabetic population. This initiative seeks to provide theoretical foundations and practical support for primary prevention strategies targeting other chronic diseases and at-risk cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for prediabetes: ①impaired fasting glucose (IFG): 6.1 mmol/L ≤ fasting plasma glucose (FPG) < 7.0 mmol/L and 2 h plasma glucose (2-hPG) after a 75 g oral glucose tolerance test (OGTT) < 7.80 mmol/L and impaired glucose tolerance (IGT): FPG<7.0 mmol/L and 7.8 mmol/L ≤ 2 hPG OGTT < 11.1 mmol/L], or HbA1c: 5.7-6.4%;
* Age ≥18 years;
* Clear awareness and comprehension ability;
* Able to use a smartphone and have access to internet at home;
* Willing to participate and sign the informed consent;
* Understand the purpose, procedure and nature of the study.

Exclusion Criteria:

* Severe cognitive impairment or mental disorder;
* Complicated with severe malignant tumours;
* Complicated with severe acute or chronic complications such as blindness, heart failure and end-stage renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Physical activity | From enrolment to the conclusion of the study, 2 weeks.
  Participants self-reported their daily physical activity levels, with the International Physical Activity Questionnaire (IPAQ) used to assess the frequency, duration, and intensity (i.e., light, moderate, and vigorous activities) of physical activity across different domains (work, transportation, household, and leisure) over the past 7 days.
Diet | From enrolment to the conclusion of the study, 2 weeks.
  Participants self-reported their daily meal consumption through periodic 24-hour dietary recalls or food diaries. These data were then used to calculate the Planetary Health Diet Score, providing a weekly assessment of diet quality.
Fasting blood glucose | From enrolment to the conclusion of the study, 2 weeks.
Two-hour postprandial blood glucose | From enrolment to the conclusion of the study, 2 weeks.
Task Completion Rate | From enrolment to the conclusion of the study, 2 weeks.
  Task Completion Rate is defined as the percentage of target users who successfully met the task criteria within the specified time frame and user scope. It directly reflects the implementation efficiency of the intervention and user adherence (e.g., dietary logging rate, exercise plan execution rate).
  Formula: Task Completion Rate = (Number of users who successfully completed the task / Total number of target users) × 100%.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | From enrolment to the conclusion of the study, 2 weeks.
Total cholesterol | On the first day of enrolment, at the conclusion of the intervention two weeks later.
Triglycerides | On the first day of enrolment, at the conclusion of the intervention two weeks later.
High-density lipoprotein cholesterol (HDL-C) | On the first day of enrolment, at the conclusion of the intervention two weeks later.
Low-density lipoprotein cholesterol (LDL-C) | On the first day of enrolment, at the conclusion of the intervention two weeks later.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China